CLINICAL TRIAL: NCT04409665
Title: The Use of Sedation Drugs in the Procedure of Administering Surfactant Without Intubation (LISA/MIST): a Randomized Study Comparing Intravenous Ketamine With Sublingual 30% Glucose
Brief Title: The Use of Sedation Drugs in the Procedure of Administering Surfactant Without Intubation (LISA/MIST)
Acronym: LISA KGS
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, PAWEL KRAJEWSKI, MD, Head of the division of neonatology, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LISA KGS TRIAL 2020
Record Dates: First submitted 2020-05-20; First posted 2020-06-01 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Neonatal Respiratory Distress Syndrome; Gestational Age Conditions
Keywords: LISA; LISA sedation; MIST; MIST sedation; Ketamine; Glucose; RDS; Newborn
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn | interventions — Ketamine; Glucose

STUDY DESIGN:
Intervention Model Description: 60 infants randomized 1:1 to receive ketamine or glucose
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketamine sedated group (Experimental): 30 randomized patients will receive Ketamine 1 mg/kg , I.V. 2 minutes before LISA
  Interventions: Drug: Ketamine
- Glucose sedated group (Active Comparator): 30 patients will receive Glucose 30% 1 mL, sublingually, 2 minutes before LISA
  Interventions: Drug: Glucose

INTERVENTIONS:
Drug: Ketamine — Patient will be sedated using Ketamine 2 minutes before the LISA procedure. 10 minutes prior the procedure and during the procedure the patient's pain and/or discomfort will be evaluated using COMFORT and FANS scales
  Arms: Ketamine sedated group
Drug: Glucose — Patient will be sedated using Glucose 2 minutes before the LISA procedure. 10 minutes prior the procedure and during the procedure the patient's pain and/or discomfort will be evaluated using COMFORT and FANS scales
  Arms: Glucose sedated group

SUMMARY:
The purpose of this study is to evaluate the efficacy and impact of intravenous ketamine or sublingual 30% glucose as sedation drugs used in preterm premature babies during the LISA procedure. The second goal is to compare the frequency of complications during LISA with both premedication regimens.

DETAILED DESCRIPTION:
All infants fulfilling the inclusion criteria during the 12 months recruitment window will potentially be enrolled in this randomized controlled trial of LISA premedication. Written informed consent will be acquired from parents or legal guardians. After the consent, infants needing the LISA will receive premedication as follows: caffeine citrate according to the clinical routine at study site, and randomly, either ketamine or sublingual glucose 30%. This study is a pilot study and 60 patients that will be randomized 1:1. Ketamine will be given in slow intravenous injection over 60 seconds. Glucose 30% will be given sublingually in the volume of 1 mL. After two minutes (from the end of administration of the study drug or reference drug), laryngoscopy will be started. To assess the effectiveness of both types of sedation, patients will be assessed using two pain assessment scales - the COMFORT scale and the FANS scale. 10 minutes before the procedure, the first assessment in the COMFORT and FANS scales will take place. The next assessment on both scales will take place during the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Infant with established Respiratory Distress Syndrome (RDS) or at risk for RDS
* Gestational age 28 0/7 - 32 6/7 weeks
* Non-invasive respiratory support with nasal CPAP (incl. BiPAP) or NIPPV
* Need for administration of exogenous surfactant

Exclusion Criteria:

* Need for intubation and mechanical ventilation at the Delivery Room
* Infant with clinically significant maxillo-facial, tracheal or pulmonary malformations

Ages: 1 Minute to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of patient sedation | First assessment 10 minutes before procedure, second during the procedure
  Assessment of patient sedation change before and after LISA using COMFORT scale
Assessment of patient sedation | First assessment 10 minutes before procedure, second during the procedure
  Assessment of patient sedation change before and after LISA using FANS scale
Comparing ketamine and glucose | Comparing the scores through study completion, an average of two years
  Comparison of the effectiveness of sedation with ketamine and glucose using the FANS scale scores. The FANS scale ranges from 0 points at minimum to 10 points at maximum. The higher the score, the lower the sedation.
Comparing ketamine and glucose | Comparing the scores through study completion, an average of two years
  Comparison of the effectiveness of sedation with ketamine and glucose using the COMFORT scale scores. The Comfort scale ranges from 8 points at minimum, to 40 at maximum. The higher the score, the lower the sedation level.

SECONDARY OUTCOMES:
Frequency of complications | During the procedure
  Monitoring the possible side effects of used drugs

CONTACTS AND LOCATIONS:
Overall Officials: Paweł Krajewski, MD, PhD, Principal Investigator — Medical University of Warsaw
Locations (1):
- Uniwersyteckie Centrum Zdrowia Kobiety Noworodka, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial will be available, after de-identification. The study protocol will also be available. These documents will be accessible to anyone who provides a methodologically sound proposal immediately following publication with no end date.
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.
Access Criteria: Anyone who provides a methodologically sound proposal.

REFERENCES:
- [Background] McPherson C, Grunau RE. Neonatal pain control and neurologic effects of anesthetics and sedatives in preterm infants. Clin Perinatol. 2014 Mar;41(1):209-27. doi: 10.1016/j.clp.2013.10.002. Epub 2013 Dec 17. PMID 24524456
- [Background] Kurepa D, Perveen S, Lipener Y, Kakkilaya V. The use of less invasive surfactant administration (LISA) in the United States with review of the literature. J Perinatol. 2019 Mar;39(3):426-432. doi: 10.1038/s41372-018-0302-9. Epub 2019 Jan 11. PMID 30635595
- [Background] Bourgoin L, Caeymaex L, Decobert F, Jung C, Danan C, Durrmeyer X. Administering atropine and ketamine before less invasive surfactant administration resulted in low pain scores in a prospective study of premature neonates. Acta Paediatr. 2018 Jul;107(7):1184-1190. doi: 10.1111/apa.14317. Epub 2018 Apr 16. PMID 29532502
- [Background] Dekker J, Lopriore E, Rijken M, Rijntjes-Jacobs E, Smits-Wintjens V, Te Pas A. Sedation during Minimal Invasive Surfactant Therapy in Preterm Infants. Neonatology. 2016;109(4):308-13. doi: 10.1159/000443823. Epub 2016 Feb 24. PMID 26907795
- [Background] McPherson C, Inder T. Perinatal and neonatal use of sedation and analgesia. Semin Fetal Neonatal Med. 2017 Oct;22(5):314-320. doi: 10.1016/j.siny.2017.07.007. Epub 2017 Jul 19. PMID 28734732
- [Background] Allegaert K, van den Anker JN. Neonatal pain management: still in search for the Holy Grail. Int J Clin Pharmacol Ther. 2016 Jul;54(7):514-23. doi: 10.5414/CP202561. PMID 27087155
- [Background] Fernandez C, Boix H, Camba F, Comunas JJ, Castillo F. Less Invasive Surfactant Administration in Spain: A Survey Regarding Its Practice, the Target Population, and Premedication Use. Am J Perinatol. 2020 Feb;37(3):277-280. doi: 10.1055/s-0039-1678534. Epub 2019 Feb 4. PMID 30716788
- [Background] Barrington K. Premedication for endotracheal intubation in the newborn infant. Paediatr Child Health. 2011 Mar;16(3):159-71. doi: 10.1093/pch/16.3.159. PMID 22379381
- [Background] Milesi C, Cambonie G, Jacquot A, Barbotte E, Mesnage R, Masson F, Pidoux O, Ferragu F, Thevenot P, Mariette JB, Picaud JC. Validation of a neonatal pain scale adapted to the new practices in caring for preterm newborns. Arch Dis Child Fetal Neonatal Ed. 2010 Jul;95(4):F263-6. doi: 10.1136/adc.2008.144758. Epub 2009 Feb 16. PMID 19221401